CLINICAL TRIAL: NCT00437463
Title: Treatment of Early Immunoglobulin A Nephropathy by ACE Inhibitor - a Randomized Controlled Trial
Brief Title: Treatment of Immunoglobulin A (IgA) Nephropathy by Angiotensin-Converting Enzyme (ACE) Inhibitor
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Trial Transparency Team, sanofi-aventis
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HOE498_6015
Record Dates: First submitted 2007-02-20; First posted 2007-02-21 (Estimated); Last update posted 2010-11-18 (Estimated); Status verified 2010-11

CONDITIONS: Glomerulonephritis
MeSH Terms: conditions — Glomerulonephritis | interventions — Ramipril

ARMS (2):
- 1 (Experimental): Ramipril
  Interventions: Drug: Ramipril
- 2 (No Intervention)

INTERVENTIONS:
Drug: Ramipril — 2.5mg and increase to 5mg if patient do not develop symptomatic hypotension
  Arms: 1

SUMMARY:
To evaluate the efficacy of the ACE inhibitor ramipril in the treatment of early IgA nephropathy.

ELIGIBILITY:
Inclusion Criteria:

* biopsy-confirmed IgA nephropathy
* proteinuria less than 0.5 g per day, normal blood pressure, and serum creatinine below 120 µmol/l

Exclusion Criteria:

* pregnant or nursing mother, or women of childbearing potential without an effective method of birth control
* history of myocardial infarction, congestive heart failure, or any other medical indication that necessitate the use of ACE inhibitor
* evidence of clinically significant hepatic, gastrointestinal, autoimmune disease
* history of malignancy, drug or alcohol abuse
* participation in any previous trial on ACE inhibitor
* taking other investigational drugs within the past 30 days
* known history of sensitivity / allergy to ACE inhibitor

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2004-07; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Development of hypertension (defined as blood pressure above 140/90 mm Hg and require anti-hypertensive therapy) | From the beginning to the end of the study
Development of proteinuria | From the beginning to the end of the study
20% decline in creatinine clearance, as determined by 24-hour urine collection or estimated by the Gault-Cockroft equation | From the beginning to the end of the study
body weight, blood pressure, pulse | From the beginning to the end of the study
Adverse effects of treatment | From the beginning to the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Yuen, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Hong Kong, Hong Kong